CLINICAL TRIAL: NCT00929266
Title: First Pilot Study Evaluating the Life Span of Autologous Cultured Red Blood Cells (cRBC) Generated From Peripheral Stem Cells in Three Healthy Volunteers - Feasibility Study
Brief Title: Cultured Red Blood Cells : Life Span in Vivo Study
Acronym: GRc2008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-AO0625-50
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers
Keywords: peripheral stem cells (PSC) donors; cultured red blood cells; In vivo half life
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The choice of conducting the study in healthy volunteers and not in patients is based on the necessity to have a healthy physiological context avoiding any situation which could lead to hemolysis. As the protocol requires mobilization with a growth factor, the donors of peripheral stem cells (PSC) receive G-CSF.
  Direct intravenous injection of labeled cRBC in a volume of 1 mL will be administered to the subjects.
  Interventions: Biological: intravenous injection of labeled cRBC

INTERVENTIONS:
Biological: intravenous injection of labeled cRBC — This step will take place within 2 months after stem cell collection. Direct intravenous injection of labeled cRBC in a volume of 1 mL, in a room reserved for the administration of radioactive drugs, situated in the nuclear medicine clinic and adjacent to the preparation laboratory, for regulatory reasons.

SUMMARY:
To study the in vivo life span in healthy volunteers of red blood cells generated in vitro from autologous peripheral stem cells. The study will be carried out in 4 phases :

* production in vitro of the equivalent of 1 ml of blood, i.e. 5x10e9 enucleated RBC from mononuclear cells isolated from an HSC graft obtained from a healthy volunteers donor.
* labeling of these cRBC with 51 Cr
* reinjection of the autologous cRBC
* follow up of the receivers for a maximum 33 days to measure the half-life span of the injected cells.

DETAILED DESCRIPTION:
1. GENERALITIES

   1.1 Clinical grade production of cRBC In this study the cRBC is both the active principle and the final product subjected to radioactive chromium labeling.

   The quantity of 5x109 cRBC to be reinjected is determined by the necessity to have a quantity of radioactivity lying between 2500 and 5000 kBq in order to have sufficient sensitivity to measure the life span.

   1.2 Hypothesis tested Since the cRBC have in vitro all the functional characteristics of native RBC, it is hypothesized that they will be viable in vivo.

   This viability will be evaluated by measuring their life span. It will be compared to the reported life span of native RBC, i.e. 30+3 days.
2. OBJECTIVES OF THE STUDY

   2.1 Principal objective Study of the life span in vivo of cultured Red Blood Cells.

   2.2 Evaluation criteria

   2.2.1 Principal: The principal criterion is the measured life span of the cRBC. It will be compared to the reported life span of native RBC, i.e. 30+3 days.

   The study involves labeling a cohort of cRBC: after administration, this cohort of cRBC will age in the circulating blood and then disappear at the end of its "life span". The results will be interpreted in the following manner:

   - if the radioactivity of the first 3 blood samples remains constant (after correction for decay), this will be taken as evidence in favor of an absence of premature cell destruction.

   The following 3 samples will be drawn later [within the limit of 30 days, after which measurement of the radioactivity of the samples will no longer be possible due to the decay of chromium 51, elimination of chromium from the cells at the rate of 1.2% per day and lack of precision of the radioactive count for very low activities]. One will conclude that the life span of the cRBC is superior to 33 days.

   - if, in the first 3 samples, the radioactivity diminishes in a significant manner and earlier than on the reference curves, three other samples taken close together will enable estimation of the mean life span of the cRBC.
3. EXPERIMENTAL PLAN

   3.1 Type of study Clinical feasibility assay.

   3.2 Experimental plan

   The study will be carried out in 4 phases:
   1. production in vitro of the equivalent of 1mL of blood, i.e. 5x109 enucleated RBC, from mononuclear cells isolated from an HSC graft obtained from a healthy benevolent donor,
   2. labeling of these cRBC with 51Cr, according to the classical protocol used to study the life span of red blood cells,
   3. reinjection of the autologous cRBC into the same donor,
   4. follow-up of the receiver for a maximal duration of 33 days to measure the half-life of the injected cells.
4. CHARACTERISTICS OF THE RECEIVERS 4.1 Description of the study population The choice of conducting the study in healthy volunteers and not in patients is based on the necessity to have a healthy physiological context avoiding any situation which could lead to hemolysis. As the protocol requires mobilization with a growth factor, the donors of peripheral stem cells (PSC) receive G-CSF.

The voluntary receivers will be recruited among intra-familial donors of PSC, in order to avoid the unnecessary exposure of a healthy donor to G-CSF.

In the context of the mobilization of HSC, they will receive for 5 days subcutaneous injections of G-CSF at a dose of 10 µg/kg body weight.

4.1.1 Collection of mononuclear cells by cytapheresis

Characteristics of the starting material:

Peripheral blood hematopoietic stem cells will not be taken for the production of cultured RBC unless the graft destined for the patient contains > 7x106 CD34+ cells/kg body weight of the patient receiver, the cell dose established in the literature as being sufficient to reconstitute the hematopoiesis of a patient receiving an allogenic graft. Thus the research protocol will incur no loss of chance for the patient.

4.1.2 Isolation of CD34+ cells for the protocol The CD34+ cells to be used for research will be selected on a positive immunomagnetic selection column using an Isolex® system. A minimum of 45x106 CD34+ cells is necessary for good functioning of the system. These limiting factors oblige us to use as starting material stem cells mobilized with G-CSF. After removal of this sample for the study, the graft will have to contain a minimum of 7x106 CD34+ cells/kg body weight of the patient.

The post-selection starting material will consist of clinical grade CD34+ cells purified by immunomagnetic selection. A purity of more than 50% CD34+ cells should be obtained after immunomagnetic selection. The percentage of viable cells will be determined by staining with trypan blue. The purified CD34+ cells will be frozen in a 4% albumin solution containing 10% DMSO and conditioned in 2.5 mL cryotubes containing 1x106 CD34+ cells. After thawing, the cell viability should be more than 50%.

A minimum of 1 million viable CD34+ cells is necessary for seeding in culture on day 0.

4.1.3 Biological characterization of the cRBC

The active principle is filtered cRBC and the final product cRBC labeled with 51Cr. As the product should be reinjected immediately after labeling, characterization will be performed on the active principle and will involve the following elements:

The active principle should consist of:

1. RBC characterized by:

   * their morphology (on slides stained with May-Grunwald-Giemsa),
   * their hemoglobin content (MHC > 25 pg measured in a Sysmex XE-2100 automate) (see 3.2.S.4.3);
2. acidophilic erythroblasts < 1.2% (in > 10,000 cells counted on a slide);
3. to the exclusion of all other cell types in > 10,000 cells counted on a slide.

4.1.4 Sufficient criteria of the active principle (cRBC)

The product will be labeled with chromium if it presents the following characteristics:

* 5 to 10x109 RBC with MHC > 25 pg,
* < 1.2% acidophilic erythroblasts,
* an absence of leukocytes. The remaining microbiological controls will be known a posteriori.

4.1.5 Labeling with chromium 51

This step will be performed in the nuclear medicine clinic. Labeling is carried out:

* using a suspension of cRBC,
* and a sterile solution of [51Cr] sodium chromate having an activity of 37 MBq/mL on calibration.

The labeling procedure itself is performed under clinically sterile conditions. The suspension is injected in 0.3 mL fractions (constraint linked to measurement of the 51Cr activity of the syringes before injection) using 2 mL syringes closed with a stopper. The maximal volume reinjected will be 5 mL by intravenous route.

4.1.6 Sufficient criteria of the final product labeled with 51Cr

The labeled product will be injected into the healthy volunteer if it presents the following characteristics:

* 51Cr activity between 2,500 KBq (minimum) and 5,000 KBq (maximum),
* an absence of 51Cr not bound to cells.

4.1.7 Injection into receivers This step will take place within 2 months after stem cell collection. Direct intravenous injection of labeled cRBC in a volume of 1 mL, in a room reserved for the administration of radioactive drugs, situated in the nuclear medicine clinic and adjacent to the preparation laboratory, for regulatory reasons.

Maintenance of a venous route until the end of the period of surveillance. Collection of 2 samples of 10 mL of blood into EDTA by venous puncture at the bend of the elbow, at T+1h and T+3h after injection.

Criteria for discharge from the clinic: absence of fever or shivering, normal blood pressure and normal clinical examination.

Total duration of the post-injection surveillance: 4 hours.

4.2 Planning of the appointments for measurement of the life span of cRBC Collection of 10 mL samples by venous puncture at the bend of the elbow and follow-up of the receivers will be carried out at the CIC St Antoine.

Transfer of the tubes to the nuclear medicine clinic.

* The third sample will be taken T+24h after injection.
* The following 3 will be taken on days chosen according to the decay estimated from the first samples (between T+48h and T+30 days after injection).

The lack of establishment of fixed dates of sampling is justified by the necessity to adapt to the kinetics of this homogenous population of cRBC, at present unknown.

A clinical examination will be carried out at each appointment. After performing the measurements, the samples will be destroyed.

In conclusion, this approach has several advantages:

1. It avoids injecting a growth factor, G-CSF, into a healthy volunteer for the sole objectives of the study.
2. The autologous situation avoids any immunological risk and any risk of transmission of infectious agents.
3. 51Cr is an emitter of gamma radiation of energy 320 keV and has a radioactive period of 27.7 days. The irradiation resulting from this study involves no measurable risk. No particular radioprotective precautions need to envisaged, either for the receiver or for those in contact with him.

ELIGIBILITY:
Inclusion Criteria:

1. Aptitude for donation of PSC validated according to the selection criteria for intra-familial donors of hematopoietic stem cells (HSC):

   * Age > 18 years and < 65 years;
   * Search by interview for risk factors pertaining to transmissible diseases;
   * Absence of significant medical antecedents;
   * Absence of severe evolutive pathology (renal, hepatic or cardiac insufficiency);
   * Serological status of the following antibodies (Ab) and antigens (Ag) determined during the 30 days preceding the donation of PSC:

     * anti-HIV 1+2 Ab (2 techniques)
     * P24 antigenemia
     * anti-HCV Ab
     * HBs Ag
     * anti-HBc Ab
     * anti-HBs Ab
     * anti-HTLV I+II Ab
     * syphilis
     * anti-CMV Ab
     * anti-toxoplasmosis Ab
     * anti-EBV Ab Determination of the blood group and search for irregular agglutinins (SIA).
2. Presence in addition of the following clinical and biological characteristics required for an assay in a healthy volunteer:

   * Results of the following biological tests within normal limits or clinically acceptable:

     * hemogram,
     * hepatic functions,
     * renal functions;
     * Absence of hemoglobinopathy on the hemoglobin electrophoresis profile;
     * Absence of G6PD or PK deficiency;
     * Absence of a radiological examination in the context of a research protocol within the last 12 months;
     * Normal arterial pressure controlled after 5 min rest in a reclining position: < 140 / 90 in three measurements at 2 min intervals;
     * ECG 12 derivations with no particularity;
     * Signature of a specific statement of informed consent to participate in the study of the life span of cRBC, in addition to the donation of HSC.

Exclusion Criteria:

* Women of child-bearing age;
* Donors carrying markers of infection: anti-HIV 1+2 Ab (2 techniques), P24 antigenemia, anti-HCV Ab, HBs Ag, anti-HTLV I+II Ab, syphilis;
* Hemoglobinopathy;
* G6PD or PK deficiency;
* Acute or chronic systemic diseases;
* Antecedents of hypersensitivity to a drug;
* Signs, symptoms or results of biological tests lying outside the limits clinically acceptable for healthy subjects;
* Known allergy to chromium.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Study of the life span in vivo of cultured Red Blood Cells. | At T+24h, T+48h and day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Antoine, Service hématologie et therapie cellulaire, Paris, France

REFERENCES:
- [Derived] Giarratana MC, Rouard H, Dumont A, Kiger L, Safeukui I, Le Pennec PY, Francois S, Trugnan G, Peyrard T, Marie T, Jolly S, Hebert N, Mazurier C, Mario N, Harmand L, Lapillonne H, Devaux JY, Douay L. Proof of principle for transfusion of in vitro-generated red blood cells. Blood. 2011 Nov 10;118(19):5071-9. doi: 10.1182/blood-2011-06-362038. Epub 2011 Sep 1. PMID 21885599
- [Derived] Abbruzzese G, Cossu G, Balocco M, Marchese R, Murgia D, Melis M, Galanello R, Barella S, Matta G, Ruffinengo U, Bonuccelli U, Forni GL. A pilot trial of deferiprone for neurodegeneration with brain iron accumulation. Haematologica. 2011 Nov;96(11):1708-11. doi: 10.3324/haematol.2011.043018. Epub 2011 Jul 26. PMID 21791473